CLINICAL TRIAL: NCT07194057
Title: "A Privacy-protecting Environment for Child Transplants Health Related and Genomic Data Integration in the European Reference Network"
Acronym: Protect_Child
Status: Not yet recruiting | Type: Observational
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Other Study IDs: PI-6796
Record Dates: First submitted 2025-08-06; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Transplant Complication; Kidney Transplant; Liver Transplant
Keywords: observational; epigenomic analysis; genomic analysis; european health data space
MeSH Terms: interventions — Whole Genome Sequencing; Epigenome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood samples will be retained for extraction of DNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Paediatric kidney and liver transplant that suffered a clinical event of interest after transplant: This cohort is made up of paediatric kidney and liver patients that had a clinical event after transplantation. The main clinical events of interest of this study are: viral infections, bacterial infections, drug-related toxicity and rejection. All patients will undergo genomic and methylomic tests to diagnose biological risk factors that could help determine the risk of developing the clinical event of interest.
  Interventions: Genetic: Whole genome sequencing; Genetic: Polygenic Risk Score Calculation; Diagnostic Test: Methylome and episignatures
- Paediatric kidney and liver transplant patients with no events after transplant: This cohort is made up of paediatric kidney and liver patients that did not develop a clinical event after transplantation. All patients will undergo genomic and methylomic tests. The genetic and methylomic results will be compared to those of the patients that developed a clinical event. The objetive is to identify biological risk factors that could help determine the risk of developing the clinical event of interest.
  Interventions: Genetic: Whole genome sequencing; Genetic: Polygenic Risk Score Calculation; Diagnostic Test: Methylome and episignatures

INTERVENTIONS:
Genetic: Whole genome sequencing — Whole genome sequencing (WGS) is an advanced genomic technique that allows for the comprehensive analysis of an individual's entire DNA sequence, including both coding and non-coding regions. In the context of pediatric transplantation, WGS offers a powerful tool for uncovering underlying genetic disorders that may influence transplant eligibility, donor-recipient compatibility, immune response, or risk of post-transplant complications. It enables the identification of rare monogenic diseases, pharmacogenomic markers relevant to immunosuppressive therapy, and potential genetic predispositions to graft rejection or infection. Integrating WGS into transplant evaluation process enhances personalized medicine approaches, contributing to improved long-term outcomes in pediatric transplant recipients.
  Other Names: Methylomic array; Polygenic risk score
Genetic: Polygenic Risk Score Calculation — A polygenic risk score (PRS) calculation will be performed to quantitatively estimate the an individual's genetic predisposition to the original disease that led to transplantation. These scores are calculated by aggregating the weighted sum of risk alleles-most commonly single nucleotide polymorphisms (SNPs)-each of which contributes a small effect size as determined by genome-wide association studies (GWAS).
Diagnostic Test: Methylome and episignatures — Methylomic analysis in paediatric transplantation refers to the comprehensive profiling and study of DNA methylation patterns across the genome to understand epigenetic modifications associated with transplant-related outcomes.
  This epigenetic approach enables the identification of differentially methylated regions (DMRs) that may correlate with clinical phenotypes, such as graft acceptance or rejection, infectious complications, or immune dysregulation.
  The studies withjin the Protect_Child_101 project will be aimed at: 1) Refinement of episignatures, to increase specificity, sensitivity and robustness of those episignatures that already exist and 2) Discovery and validation of new disease, gene or variant specific mDNA signatures.

SUMMARY:
Protect_Child_101 is an observational study to be performed in children that have undergone a liver or renal transplant.

The aim of this study is to analyse small variations in the genetic material (DNA) of transplanted children. The investigators will also study a type of chemical 'marks' called methylations, which do not change the DNA itself, but can affect how it functions. These marks can influence how certain diseases develop or how the body responds to transplantation.

Specifically, investigators seek to discover:

* Whether there are genetic or epigenetic (methylation) alterations that may explain why some children develop serious diseases that require transplantation.
* If these alterations can help us predict possible complications after transplantation, such as organ rejection, infections, organ failure, cancer development.

Within this study, data from the child's medical history will be collected. The data to be collected are demographic data (gender, age, ethnicity), clinical data, personal and family history possibly related to his/her disease, course and evolution of the disease, and complementary and laboratory examinations collected from his/her clinical history.

The only non-routine tests to be performed will be the genomic and methylomic tests. Nevertheless, these determinations will be performed on samples obtained during the child's routine care. No extra intervention is planned as part of this study.

Samples and clinical data will be collected at different time points after transplantation. Schematically, collection is planned for months 0, 1, 3, 6, 12 and 24 post-transplant. In addition to these pre-established points, comprehensive data collection will be attempted when the child suffers a relevant clinical event, e.g. infection, treatment toxicity, organ rejection (post-transplant complication).

ELIGIBILITY:
Inclusion Criteria:

* ● Paediatric patients (6 months to 18 years old) with liver or kidney transplant.

Both patients with de novo transplantation or in follow-up can be included in the study.

* For the retrospective cohort, only patients within the first 5 years after transplantation will be included.
* Patients and/or parents agreeing to participate in the study and provide consent for the obtention of clinical data and samples for genomic and methylomic analysis and the use of the information according to the protocol.

Exclusion Criteria:

* Patients that are not being followed up in the clinical site.
* Subjects alternating between different clinical sites. Subjects/Tutors that don't understand the informed consent form.
* Subject or their legally authorized representative does not sign the informed consent document.
* Re-transplantation or AB0-incompatible transplantation.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will enroll paediatric patients that have underdone a renal i liver transplant
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Epstein Barr Infection | From transplant until end of post-transplant follow-up period (up to 7years)
  Number of Espstein Barr infections defined as >3500 copies in PCR in peripheral blood
Cytomegalovirus infection | From transplant until end of post-transplant follow-up period (up to 7 years)
  A) Primary CMV infection after transplant with or without CMV disease (>1000 copies/ml in peripheral blood in patients with previous negative CMV serology) B) Secondary CMV infection after transplant (any PCR with CMV disease or CMV >1000 copies/ml in asymptomatic patients)
BK virus infection | From transplant until end of post-transplant follow-up period (up to 7 years)
  Positive BK viremia (define cut-off level) and/or histological evidence of BK nephropathy
Cholangitis | From transplant until end of post-transplant follow-up period
  Worsening of liver function tests accompanied by an elevation in inflammatory markers, with or without a positive blood or bile culture.
Urinary Tract Infection | From transplant until end of post-transplant follow-up period (up to 7 years)
  Positive urine cultures AND increased inflammation marker (e.g. CRP) or fever
Sepsis | From transplant until end of post-transplant follow-up period (up to 7 years)
  SIRS in relation to infectious cause +/- positive blood cultures
Renal Calcineurin Inhibitors toxicity | From transplant until end of post-transplant follow-up period (up to 7 years)
  Histological evidence of kidney CNI-related kidney damage
Mycophenolate mofetil toxicity | From transplant until end of post-transplant follow-up period (up to 7 years)
  Evidence of myelosuppression during therapy without any other proven cause and/or Clinical/histological evidence of MMF-related enteropathy
mTOR inhibitor toxicity | From transplant until end of post-transplant follow-up period (up to 7 years)
  mTOR induced-proteinuria (occurrence of proteinuria after mTOR exposure with resolution after treatment suspension)
Thrombotic microangiopathy | From transplant until end of post-transplant follow-up period (up to 7 years)
  Ocurrence of no non immune-mediated hemolytic anemia and/or thrombocytopenia and/or hypertension and/or proteinuria with histological evidence of kidney TMA
Kidney rejection episode | From transplant until end of post-transplant follow-up period (up to 7 years)
  Histological evidence based on Banff criteria
Liver rejection episode | From transplant until end of post-transplant follow-up period (up to 7 years)
  Histological evidence based on Banff criteria
Chronic liver rejection | From transplant until end of post-transplant follow-up period (up to 7 years)
  Histological evidence based on Banff criteria
Chronic kidney rejection | From transplant until end of post-transplant follow-up period (up to 7 years)
  Histological evidence based on Banff criteria
Chronic renal failure after pLTx | From transplant until end of post-transplant follow up period (up to 7 years)
  Elevation of serum-creatinine for 3>months
Chronic liver failure (graft chirrosis and fibrosis) | From transplant until end of post-transplant follow up period (up to 7 years)
  Ocurrence of portal hypertension diagnosis both clinical (ascites, splenomegaly, varices) and analytical (thrombocytopenia) presentation.

SECONDARY OUTCOMES:
Liver Primary non-function | From transplant to post-trasnplant follow-up period (up to 7 years)
  Requirement for immediate re-transplantation
Liver Primary non-function | From transplant to post-transplant follow-up period (up to 7 years)
  Early death within the first 7 or 14 days following LT after exclusion of other identifiable causes of graft function such as vascular complications, rejection, or infection
Liver Primary non-function | From transplant to post-trasnplant follow-up period (up to 7 years)
  Ocurrence of at least 2 of the following within 7 days post-transplant:
  * Alanine aminotransferase (ALT) greater than or equal to 2,000 U/L
  * INR greater than or equal to 10 mg/dl
  * Acidosis (Defined as one of the following: a) Arterial PH less or equal to 7,30. b) Venous pH less than or equal to 7,25. c) Lactate greater than or equal to 4 mmol/L)
Kidney primary non-function | From transplant until end of post-transplant follow-up period (up to 7 years)
  Persistence of dialysis status or eGFR <15 ml/min/1.7 m2
Liver early allograft dysfunction | From transplant until end of post-transplant follow-up period (up to 7 years)
  One of the following laboratory criteria within the 7 first days post transplant:
  * Serum bilirubin ≥10 mg/dL (171 μmol/L) on day 7
  * INR ≥1.6 on day 7
  * AST or ALT >2000 IU/L within the first 7 days.
  Or, for 5 consecutive days after day 7:
  * Bilirubin > 10 mg/ dL
  * INR > 1.6
  * Serum Urea > 100 mg/dL
Delayed kidney Graft Function | From transplant until end of post-transplant follow-up period (up to 7 years)
  Need for dialysis within the first 7 days after kidney transplantation
Vascular Complications | From transplant until end of post-transplant follow-up period (Up to 7 years)
  Hepatic artery thrombosis (HAT) or portal vein stenosis (may lead to ischemic injury and chronic dysfunction)
Biliary Complications | From transplant until end of post-transplant follow-up period (up to 7 years)
  Biliary structures, leaks, or ischemic cholangiopathy due to vascular insufficiency can cause chronic dysfunction.
Urological complications | From transplant until end of post-transplant follow-up period (up to 7 years)
  Need of re-intervention due to post-surgical events
Post-transplant lymphoproliferative disease | From transplant until end of post-transplant follow-up period (up to 7 years)
  Histological diagnosis of PTLD: histology, immunohistochemistry, EBV detection (EBER in situ hybridization), and clonality studies, classified according to WHO PTLD categories.
Post-transplant lymphoproliferative disease | From transplant until end of post-transplant follow-up period (up to 7 years)
  Radiological diagnosis of PTLD: heterogeneous extranodal masses, allograft involvement, and CNS or visceral lesions.
Diabetes | From transplant until end of post-transplant follow-up period (up to 7 years)
  The diagnosis is confirmed when one of the following criteria is met on two separate occasions:
  Fasting plasma glucose (FPG): ≥126 mg/dL (7.0 mmol/L) after at least 8 hours fasting.
  Oral glucose tolerance test (OGTT): 2-hour plasma glucose ≥200 mg/dL (11.1 mmol/L) after a 75 g oral glucose load.
  Hemoglobin A1c (HbA1c): ≥6.5%, using a standardized assay.
  Random plasma glucose: ≥200 mg/dL (11.1 mmol/L) in the presence of classic symptoms of hyperglycemia (polyuria, polydipsia, weight loss).
Posterior reversible encelopathy (PRES) | From transplant until end of post-transplant follow-up period (up to 7 years)
  Ocurrence of acute neurologic symptoms (headache, seizures, altered consciousness or visual disturbances) with typical neuroimaging (CT, MRI) findings (bilateral areas of white matter edema in the posterior cerebral hemispheres).
Mortality | From transplant until end of post-transplant follow-up period (up to 7 years)
  Death by any cause
Relapse of primary immune mediated disease | From transplant until end of post-transplant follow-up period (up to 7 years)
  Ocurrence of nephrotic range proteinuria after kidney transplant (excluding other causes)
Relapse of primary immune mediated disease | From transplant until end of post-transplant follow-up period (up to 7 years)
  histological findings of Focal segmental glomerulosclerosis (FSGS) in kidney biopsy in a patient with primary FSGS
Graft survival | From transplant until end of post-transplant follow-up period (up 7 years)
  Time from transplant to the need for dialysis or entry onto the re- transplant list.

CONTACTS AND LOCATIONS:
Locations (4):
- University Medical Center Hamburg-Eppendorf (UKE),, Hamburg, Germany
- Italy (2):
  - Mediterranean Institute for Transplantation (ISMETT), Palermo, Sicily
  - University Hospital Padova, Padua
- Hospital Universitario La Paz, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No